CLINICAL TRIAL: NCT00534898
Title: Comparison Efficacy of Bexarotene and Fenretinide as Addition to Antipsychotic Treatment in Schizophrenia Patients: Double-blind Placebo Controlled Study
Brief Title: Bexarotene and Fenretinide as Addition to Antipsychotic Treatment in Schizophrenia Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study withdrawn due to lack financial support
Sponsor: Beersheva Mental Health Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LMR250850MHC
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2007-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Cognition
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Bexarotene; Fenretinide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Bexarotene
Drug: Fenretinide
Drug: Placebo

SUMMARY:
Background: In this proposed study, we aim to investigate safety and efficacy of two synthetic retinoids - bexarotene (Targretin; LGD1069; 4-[1-{5,6,7,8-tetrahydro-3,5,5,8,8-pentamethyl-2-naphthalenyl} ethenyl] benzoic acid) and fenretinide (Dihydroceramide N-(4-Hydroxyphenyl retinamide) on severity of psychopathology and cognitive impairment in schizophrenia patients in an double-blind, placebo-controlled study. The rationale behind add-on these medications to ongoing antipsychotic treatment in schizophrenia patients is based on both the retinoid dysregulation hypothesis: the growth factors deficiency and synaptic destabilization hypothesis of schizophrenia. Furthermore, in our preliminary open clinical trial, we found that a low dose of bexarotene (Targretin, 75 mg/day) was safe and led to significant improvement on total PANSS scores, general psychopathology, on the positive and the dysphoric mood factor scores. The aim of the present study was to provide further insight into the safety and efficacy of bexarotene in comparison to fenretinide (a medication with smaller potential of adverse effects) and placebo in patients suffered from schizophrenia.

DETAILED DESCRIPTION:
In this clinical trial, a minimal dose of bexarotene (Targretin, 75 mg/day) or fenretinide 5 mg/day or placebo will be added for 8 weeks to the stable ongoing antipsychotic treatment of 90 schizophrenia patients. Participants will be assessed at baseline and after 2, 4 and 8 weeks of treatment. A battery of research instruments will be used for assessment of efficacy and safety (psychopathology, and side effects). In addition, cholesterol and triglyceride levels, liver and thyroid function tests and a blood cell count will be monitored at baseline and during therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years, male or female
2. DSM-IV criteria for schizophrenia
3. Ability and willingness to sign informed consent for participation in the study
4. Stable blood parameters
5. Only patients who had a normal baseline fasting triglyceride

Exclusion criteria:

1. Lipid abnormalities.
2. Leukopenia or neutropenia.
3. Evidence of organic brain damage, mental retardation, alcohol or drug abuse
4. Renal disease
5. Hepatic dysfunction.
6. A history of pancreatitis.
7. Thyroid axis alterations
8. Suicide attempt in past year.
9. Cataracts.
10. High dose of vitamin A daily treatment.
11. Patients with a known hypersensitivity to bexarotene or other components of the product.
12. Pregnant women or a woman who intends to become pregnant.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Lerner, MD, PhD, Principal Investigator — Ben-Gurion University of the Negev; Chanoch Miodownik, MD, Study Director — Ben-Gurion University of the Negev
Locations (1):
- Be'er Sheva Mental Health Center, Sha'ar Menashe Mental Health Center, Be'er Sheva, Hadera, Israel